CLINICAL TRIAL: NCT04050293
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter, Parallel Group Study to Evaluate the Efficacy and Safety of SPN-538 as a Therapy for the Prevention of Migraine in Subjects Ages 6-11 Years
Brief Title: Therapy for Migraine Prevention in Children 6-11 Years of Age
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulty in recruitment
Sponsor: Supernus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 538P401
Record Dates: First submitted 2019-08-02; First posted 2019-08-08 (Actual); Results first posted 2025-11-21 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-12

CONDITIONS: Migraine Disorders; Headache Disorders
MeSH Terms: conditions — Migraine Disorders; Headache Disorders

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized, placebo-controlled, 2-arm, parallel group study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SPN-538 (Topiramate XR capsule) (Experimental): Participants will be treated with SPN-538
  Interventions: Drug: SPN-538
- Placebo (Placebo Comparator): Participants will be treated with Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SPN-538 — Participants will receive SPN-538
  Arms: SPN-538 (Topiramate XR capsule)
Drug: Placebo — Participants will receive Placebo
  Arms: Placebo

SUMMARY:
The aim of this study is to evaluate the effect of SPN-538 for the prophylaxis of migraine in pediatric patients 6 to 11 years old.

DETAILED DESCRIPTION:
The study is to assess the efficacy and safety of SPN-538 in reducing the monthly migraine headache frequency in pediatric patients with migraine.

This is a multicenter, randomized, double-blind, placebo-controlled, 2-arm, parallel group Phase 4 study in children 6 to 11 years of age to evaluate the efficacy and safety of SPN-538 for the prevention of migraine. SPN-538 (or matching placebo) will be administered as a single oral dose once a day (QD), starting at 25 mg/day and increasing every 2 weeks in 25 mg increments to a target dose of 2 to 3 mg/kg/day or the maximum tolerated dose (MTD), whichever is less. The total study duration is a maximum of 34 weeks including a Screening Period, Prospective Baseline Period of up to 8 weeks, a Treatment Phase of 20 weeks (8 weeks titration followed by 12 weeks of maintenance dosing), a Dose Tapering Period of 1 to 3 weeks, and a Safety Follow-up Period of 1 to 3 weeks

ELIGIBILITY:
Inclusion Criteria:

* Otherwise, healthy male or female (6 to 11 years of age at the time of screening) with a history of migraine with or without aura for at least 6 months prior to screening, 3-12 migraine episodes and no more than 14 headache days (migraine and non-migraine) per month during the 3 months prior to Screening and during the 28-day Prospective Baseline Period, a PedMIDAS Disability score of ≥20 and ≤139 and weight at least 20 kg and no more than 60 kg.

Exclusion Criteria:

* Subjects with chronic migraine (>14 headache days per month), cluster headaches, or migraine aura without headache and who are unable to distinguish migraines from other headache types.
* Subjects with more than 14 headache days during the 28-day Prospective Baseline Period
* Have taken any disallowed migraine preventive medication including TPM within 14 days prior to the start of the Prospective Baseline Period; or used onabotulinumtoxinA (Botox®) within 3 months prior to Screening.
* Failure to respond to topiramate prophylaxis therapy (2 to 3 mg/kg/day) for a minimum of 3 months, or those who have previously discontinued TPM due to AEs within 6 months prior to Screening.
* Failure to more than 2 adequate clinical trials of an established prophylactic antimigraine regimen within 6 months prior to Screening.
* Current use of antipsychotics, antimanics, barbiturates, benzodiazepines amitriptyline, lithium, valproic acid, tricyclic antidepressants, AEDs, calcium channel blockers, sedatives, SSRIs, NSRIs, CGRP receptor antagonists, CBD oil, herbal preparations/supplements such as feverfew or St John's wort and/or any medications that could impair or decrease thinking and concentration.
* Overuse of analgesic or migraine-specific agents for acute treatment of migraine (>10 treatment days/month of ergot-containing medications or triptans; or >15 treatment days/month with simple analgesics (including non steroidal anti-inflammatory drugs [NSAIDs]), or use of narcotics.
* Use of non-pharmacologic complementary and alternative prophylactic approaches for migraine prevention, such as neuromodulation, acupuncture, behavioral interventions, spinal manipulation, occipital nerve block and neurofeedback.
* Diagnosis of psychiatric disorder (e.g., psychosis, bipolar disorder, major depression, generalized anxiety disorders), or documented developmental delays or impairments (e.g., autism, cerebral palsy, or mental retardation).
* Subjects with seizures or a history of seizure-like events.
* Known history of visual field defects, neurological disorder or structural disorder of the brain from birth; head trauma or previous CNS surgery.
* Evidence of active suicidal ideation and/or suicidal behaviors 6 months before screening, pregnancy, active liver disease or abnormal kidney function.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2020-07-14 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gianpiera Ceresoli-Borroni, PhD, Study Director — Employee of Supernus
Locations (1):
- CNS Healthcare, Memphis, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total of 60 participants were screened for eligibility; 26 participants randomized to receive double-blind treatment.
Groups:
- Placebo: Participants received Placebo once a day.
- SPN-538: Participants received SPN-538 once a day starting at 25 mg/day and increasing every 2 weeks in 25-mg increments to a target dose of 2 to 3 mg/kg/day or the maximal tolerated dose (MTD), whichever is less.
Period: Overall Study
Arm/Group | Placebo | SPN-538
Started | 13 | 13
Completed | 10 | 11
Not Completed | 3 | 2
Not completed — Lost to Follow-up | 1 | 2
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population includes all randomized participants who received at least one dose of study medication.
Groups:
- Placebo: Patients received Placebo once a day.
- Total: Total of all reporting groups
Arm/Group | Placebo | SPN-538 | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 13 | 13 | 26
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.2 (1.59) | 8.2 (1.68) | 8.2 (1.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 9 | 15
  Male | 7 | 4 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 7 | 14
  White | 6 | 6 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 13 | 26
Baseline Migraine Frequency [Mean (Standard Deviation); unit: monthly migraine day] — Prospective baseline was defined as the non-missing value collected most recent to and before the time of the very first dose of the study medication, in the last 4 weeks before randomization. The tool for collecting daily information about headaches was the Headache Diary - Preventive Therapies. A similar diary was used in the CHAMP study by Powers et al (Powers et al., 2017). The Headache Diary was presented in an electronic format uploaded on a dedicated electronic patient reported outcome (ePRO) data collection application; a device was provided as needed. Population: The measure is the 28-day rate for the prospective baseline defined as the total number of migraine days during the last 4 weeks prior to randomization/total number of days with non-missing headache data during the 28 days prior to randomization *28 in the FAS population.
  Number of participants is from the FAS: participants who received at least one dose of study medication and have a baseline and at least one valid post-baseline assessment of monthly migraine based on the headache diary data.
  monthly migraine day
    number analyzed (Participants) | 11 | 13 | 24
    (all) | 7.22 (3.434) | 6.09 (1.365) | 6.61 (2.535)
Height [Mean (Standard Deviation); unit: centimeter] | 133.6 (10.57) | 137.5 (10.97) | 135.6 (10.74)
Weight [Mean (Standard Deviation); unit: Kilograms] | 37.2 (9.81) | 41.6 (13.29) | 39.4 (11.67)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per square meter] | 20.51 (3.564) | 21.35 (4.285) | 20.93 (3.885)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Monthly Migraine Days (MMDs) in Children 6 to 11 Years Old With Migraine.
Description: The primary efficacy endpoint was the change in rate of the MMDs relative to the Prospective Baseline Period (PBP). The 28-day rate of MMDs was calculated as the ratio of the # days of migraine during the last 4 weeks of PBP and the # days with non-missing headache record in the electronic diary during the last 4 weeks of the 20-week double-blind Treatment Phase, x 28. The primary outcome measure was recorded on headache electronic diary uploaded on a Patient Reported Outcome (ePRO) application. The electronic diary will serve as the primary tool to collect daily headaches information.
Time Frame: Baseline, Titration Period 1 (Month 1), Titration Period 2 (Month 2), Maintenance Period 1 (Month 3), Maintenance Period 2 (Month 3), Maintenance Period 2 (Month 4) and Maintenance Period 3 (Month 5)
Population: Full Analysis Set (FAS) included participants who received at least one dose of study medication and have a baseline and at least one valid post-baseline assessment of monthly migraine based on the headache diary data.
  The number of participants in some rows differs from the overall number as some participants discontinued the study before the specific time points.
Measure: Mean (Standard Deviation); unit: monthly migraine days
Arm/Group | Placebo | SPN-538
Number analyzed (Participants) | 11 | 13
monthly migraine days
  Titration Period 1 (Month 1) | -2.89 (1.919) | -3.08 (0.830)
  Titration Period 2 (Month 2): number analyzed (Participants) | 11 | 12
  Titration Period 2 (Month 2) | -4.85 (2.199) | -3.38 (2.057)
  Maintenance Period 1 (Month 3): number analyzed (Participants) | 10 | 12
  Maintenance Period 1 (Month 3) | -4.25 (2.903) | -4.35 (1.977)
  Maintenance Period 2 (Month 4): number analyzed (Participants) | 10 | 11
  Maintenance Period 2 (Month 4) | -5.41 (3.049) | -4.18 (2.279)
  Maintenance Period 3 (Month 5): number analyzed (Participants) | 10 | 11
  Maintenance Period 3 (Month 5) | -4.32 (2.477) | -4.50 (2.410)

ADVERSE EVENTS:
Time Frame: Baseline (Day 1) to Week 26
Description: Treatment Emergent Adverse Event (TEAE) is an adverse event (AE) with a start date on or after the first dose of study medication is taken, or that worsened following first administration of study medication.
Arm/Group | Placebo | SPN-538
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 4/13 | 4/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=13) | SPN-538 (N=13)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
Croup infectious (Infections and infestations) | 1 (1) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 1 (1)
Mood altered (Psychiatric disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Rhinitis allergic (Immune system disorders) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Ammonia increased (Investigations) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to study termination (difficulty in recruitment), the target number of participants needed to achieve statistically reliable results was not met.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-12-14): https://cdn.clinicaltrials.gov/large-docs/93/NCT04050293/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-06): https://cdn.clinicaltrials.gov/large-docs/93/NCT04050293/SAP_001.pdf